CLINICAL TRIAL: NCT02004444
Title: JC Virus Reactivation in Multiple Sclerosis
Acronym: JCV in MS
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Multiple Sclerosis Society (Other); Biogen (Industry)
Responsible Party: Principal Investigator, Igor Koralnik, Chief, Division of NeuroVirology, Beth Israel Deaconess Medical Center
Other Study IDs: 2010P-000249 RG 452 3-A-1
Record Dates: First submitted 2013-11-20; First posted 2013-12-09 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Progressive Multifocal Leukoencephalopathy; Multiple Sclerosis
Keywords: JC Virus; Natalizumab
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood, Urine, and Cerebrospinal Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Natalizumab 18 months: 10 patients on continuous natalizumab monotherapy for 18 months
- Natalizumab 24 months: 10 patients on continuous natalizumab monotherapy for 24 months
- Natalizumab 36 months: 10 patients on continuous natalizumab monotherapy for 36 months
- IFN-beta 36 months: 10 patients on continuous interferon-beta monotherapy for 36 months
- Untreated: 10 untreated patients

SUMMARY:
JC virus is a benign virus which infects approximately up to 90% of the normal adult population. However, it may be reactivated in people who have a decreased immune function as in HIV infection, cancer, chemotherapy, transplant recipients, or in MS patients treated with natalizumab (Tysabri). In these patients, JC virus can cause a severe brain disease called Progressive Multifocal Leukoencephalopathy (PML), for which there is no cure.

As of September 2013, 400 MS patients in the world, who have been treated with natalizumab, have developed PML. The risk of PML is approximately 5 patients in 1000 after 24 months on the drug. Researchers do not know exactly in which cells of the body the virus lives but it has been isolated from the blood, urine, cerebrospinal fluid (CSF), and from the brains of patients with immunosuppression.

In this study, the investigators wish to determine precisely where the virus lives, and how the body prevents it from causing brain disease.

Because of the association of PML with natalizumab, the investigators would like to see if there is a difference in the amounts of virus in blood, urine, and CSF found in MS patients treated with natalizumab or those treated with different medications for MS, or those not treated at all. The investigators hope that this knowledge will allow us to find better ways of preventing the development of PML as well as treatments for patients with PML.

DETAILED DESCRIPTION:
Subjects selected for participation in this study have been diagnosed with Multiple Sclerosis (MS). Of the MS patients enrolled in the study, some have been treated with natalizumab or a different medication for MS, and others have not been treated at all. All MS patients enrolled have their blood tested for the presence of the JC virus. Those testing negative for the JC virus do not continue in the study. Those testing positive for the JC virus continue participating in the study, and provide a urine sample, blood sample, lumbar puncture, and a neurological exam. Approximately 65 people will take part in this study at Beth Israel Deaconess Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Sclerosis, relapsing remitting

Exclusion Criteria:

* JCV sero-negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected mostly from the neurology clinic at Beth Israel Deaconess Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Molecular determinants of JCV reactivation in blood, urine, and CSF | 1 day
  Characterize the phenotype of the cells carrying JCV in the blood of MS patients after 18, 24 and 36 months on continuous natalizumab therapy and in interferon-beta treated and untreated MS subjects, and analyze the molecular determinants of JCV reactivation in their blood, urine and CSF.

SECONDARY OUTCOMES:
Humoral and Cellular Immune Response to JCV | 1 day
  Evaluate the humoral and cellular immune response against JCV in MS patients after 18, 24 and 36 months on continuous natalizumab therapy and in interferon-beta treated and untreated MS subjects, and correlate these findings with JCV reactivation in different compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Igor J Koralnik, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Chalkias S, Dang X, Bord E, Stein MC, Kinkel RP, Sloane JA, Donnelly M, Ionete C, Houtchens MK, Buckle GJ, Batson S, Koralnik IJ. JC virus reactivation during prolonged natalizumab monotherapy for multiple sclerosis. Ann Neurol. 2014 Jun;75(6):925-34. doi: 10.1002/ana.24148. Epub 2014 Jun 10. PMID 24687904